CLINICAL TRIAL: NCT01900535
Title: A Randomized Clinical Trial to Evaluate and Compare the Efficacy of Triphala Mouthwash With 0.2% Chlorhexidine in Hospitalized Patients With Periodontal Diseases
Brief Title: Evaluation and Comparison of the Efficacy of Triphala Mouthwash and 0.2% Chlorhexidine
Status: Completed | Type: Observational
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, Dr. Ritam S. Naik Tari, Dr., Tatyasaheb Kore Dental College
Other Study IDs: TKDC- 11
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Periodontal Disease
Keywords: chlorhexidine; gingivitis; periodontitis
MeSH Terms: conditions — Periodontal Diseases; Gingivitis; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the usefulness of triphala mouthwash in comparison with the gold standard chlorhexidine in hospitalized and periodontally diseased patients.

ELIGIBILITY:
Inclusion Criteria:

* age group of 20-65 years having periodontal diseases according to American Academy of Periodontology (AAP) classification 1999

Exclusion Criteria:

* patients seeking any periodontal treatment during the course of study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants were selected from patients admitted to three different medical hospitals namely Mahatma Gandhi Hospital, New Pargaon, Sub district Government Hospital, Kodoli and Yeshwant Chavan Hospital, Kodoli
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
plaque index | 15 days

SECONDARY OUTCOMES:
gingival index | 15 days